CLINICAL TRIAL: NCT03322423
Title: Evaluation of Two Marketed Multifocal Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CR-5860
Record Dates: First submitted 2017-09-28; First posted 2017-10-26 (Actual); Results first posted 2019-01-08 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2018-12

CONDITIONS: Visual Performance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Test 1 Multifocal/Test 2 Multifocal OR Test 2 Alternative (Active Comparator): Subjects who are habitual soft contact lens wearers, at least 40 years of age and no more than 70 years of age, will wear Test 1 Multifocal then Test 2 Multifocal OR Test 2 Alternative (based on lens optimization- subject's lens power), for approximately 8-12 days of wear with an approximately 4-8 day washout period.
  Interventions: Device: Multifocal Contact Lens 1; Device: Multifocal Contact Lens 2; Device: Spherical Contact Lens 2
- Test 2 Multifocal OR Test 2 Alternative/Test 1 Multifocal (Active Comparator): Subjects who are habitual soft contact lens wearers, at least 40 years of age and no more than 70 years of age, will wear Test 2 Multifocal OR Test 2 Alternative (based on lens optimization- subject's lens power) then Test 1 Multifocal, for approximately 8-12 days of wear with an approximately 4-8 day washout period.
  Interventions: Device: Multifocal Contact Lens 1; Device: Multifocal Contact Lens 2; Device: Spherical Contact Lens 2

INTERVENTIONS:
Device: Multifocal Contact Lens 1 — Dailies Total 1 Multifocal Contact Lens
  Other Names: Test 1 Multifocal , delefilcon A
Device: Multifocal Contact Lens 2 — Biotrue ONEday for Presbyopia Contact Lenses
  Other Names: Test 2 Multifocal, nesofilcon A
Device: Spherical Contact Lens 2 — BioTrue ONEDay Spherical
  Other Names: Test 2 Alternative, nesofilcon A

SUMMARY:
This is a single-masked, randomized, cross-over, dispensing, 6- visit pilot study. The purpose of this clinical study is to evaluate the performance of two marketed multifocal lenses.

ELIGIBILITY:
Inclusion Criteria:

* Potential subjects must satisfy all of the following criteria to be enrolled in the study:

  1. The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
  2. The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.
  3. The subject must be between at least 40 years of age and not greater than 70 years of age.
  4. The subject's distance spherical equivalent refraction must be in the range of +3.75 D to -3.75 D.
  5. The subject's refractive cylinder must be ≤ -0.75 D in each eye.
  6. The subject's ADD power must be in the range of +0.75 D to +2.50 D in each eye.
  7. The subject must have best corrected visual acuity of 20/20-3 or better in each eye.
  8. The subject must own a pair of wearable spectacles if required for their distance vision.
  9. The subject must be an adapted soft contact lens wearer in both eyes (i.e. worn lenses a minimum of 2 days per week for at least 8 hours per wear day, for 1 month or more duration).
  10. The subject must either be wearing a presbyopic contact lens correction (e.g., reading spectacles over contact lenses, multifocal or monovision contact lenses, etc.) or respond positively to at least one symptom on the "Presbyopic Symptoms Questionnaire".

      Exclusion Criteria:
* Potential subjects who meet any of the following criteria will be excluded from participating in the study:

  1. Ocular or systemic allergies or disease, or use of medication which might interfere with contact lens wear.
  2. Pregnancy or lactation.
  3. Currently diagnosed with diabetes.
  4. Infectious diseases (e.g. hepatitis, tuberculosis) or an immune-suppressive disease (e.g. HIV).
  5. Clinically significant (Grade 3 or 4) corneal edema, corneal vascularization, corneal staining, tarsal abnormalities or bulbar injection, or any other corneal or ocular abnormalities which would contraindicate contact lens wear.
  6. Entropion, ectropion, extrusions, chalazia, recurrent styes, dry eye, glaucoma, history of recurrent corneal erosions.
  7. Any previous, or planned, ocular or intraocular surgery (e.g., radial keratotomy, PRK, LASIK, lid procedures, cataract surgery, retinal surgery, etc.).
  8. A history of amblyopia, strabismus or binocular vision abnormality.
  9. Any ocular infection or inflammation.
  10. Any ocular abnormality that may interfere with contact lens wear.
  11. Use of any ocular medication, with the exception of rewetting drops.
  12. History of herpetic keratitis.
  13. Participation in any contact lens or lens care product clinical trial within 30 days prior to study enrollment.
  14. Employee of clinical site (e.g., Investigator, Coordinator, Technician)

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2017-09-11 (Actual); Primary Completion 2017-11-04 (Actual); Study Completion 2017-11-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Golden Vision, Sarasota, Florida
  - ABQ Eye Care, Albuquerque, New Mexico
  - Sacco Eye Group, Vestal, New York
  - West Bay Eye Associates, Warwick, Rhode Island
  - Botetourt Eyecare, LLC, Salem, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 78 subjects were enrolled into this study. Of the enrolled all 78 were dispensed at least one study lens. Of the dispensed subjects 71 completed the study, while 7 subjects were discontinued.
Groups:
- Delefilcon A/Nesofilcon A: All subjects that were randomized to receive the delefilcon A lens during the first period of the study and the nesofilcon A lens during the second period of the study.
- Nesofilcon A/Delefilcon A: All subjects that were randomized to receive the nesofilcon A during the first period of the study and the delefilcon A lens during the second period of the study.
Period: Period 1
Arm/Group | Delefilcon A/Nesofilcon A | Nesofilcon A/Delefilcon A
Started | 38 | 40
Completed | 36 | 38
Not Completed | 2 | 2
Not completed — Subject no longer eligible | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Incorrect Lens Dispensed | 1 | 0
Not completed — Unsatisfactory Lens Fitting | 1 | 0
Period: Period 2
Arm/Group | Delefilcon A/Nesofilcon A | Nesofilcon A/Delefilcon A
Started | 36 | 38
Completed | 35 | 36
Not Completed | 1 | 2
Not completed — Dispensed incorrect lens in left eye | 0 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Subject not eligible for Pytergiumectomy | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Dispensed Subjects: All subjects that were dispensed a study lens.
Arm/Group | All Dispensed Subjects
Number analyzed (Participants) | 78
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.9 (7.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61
  Male | 17
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 1
  Black or African American | 2
  White | 73
  American Indian or Alaska Native | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 78

OUTCOME MEASURES:

1. Primary Outcome: Distance Binocular Visual Acuity
Description: Distance visual acuity was assessed for each subject in both eyes under a high luminance high contrast condition using ETDRS (Early Treatment Diabetic Retinopathy Study) charts.
Time Frame: 1-Week Follow-up
Population: All subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: Eyes
Groups:
- Delefilcon A: All subjects that wore the delefilcon A lens during either the first or second period of the study.
- Nesofilcon A: All subjects that wore the nesofilcon A lens during either the first or second period of the study.
Arm/Group | Delefilcon A | Nesofilcon A
Number analyzed (Participants) | 65 | 65
Number analyzed (Eyes) | 110 | 110
logMAR | -0.056 (0.0842) | -0.075 (0.0759)
Statistical Analysis 1: Comparison: Delefilcon A; Test type: Superiority — Statistical superiority was concluded if the upper limit of the confidence intervals of the Test lens was below +0.01 logMAR for distance; Linear mixed model analysis; Linear mixed model using the Kenward and Roger method for the denominator degrees of freedom; Least-Square Mean Estimate = -0.058, 95% CI 2-sided [-0.080 to -0.035], Standard Error of Mean 0.0114
Statistical Analysis 2: Comparison: Nesofilcon A; Test type: Superiority — [test comment as in outcome 1, analysis 1]; Linear mixed model analysis; Linear mixed model using the Kenward and Roger method for the denominator degrees of freedom; Least-Square Mean Estimate = -0.076, 95% CI 2-sided [-0.099 to -0.054], Standard Error of Mean 0.0114

2. Primary Outcome: Near Binocular Visual Acuity
Description: Near visual acuity was assessed for each subject in both eyes under a high luminance high contrast condition using reduced Guillon-Poling Charts.
Time Frame: 1-Week Follow-up
Population: All subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: Eyes
Arm/Group | Delefilcon A | Nesofilcon A
Number analyzed (Participants) | 65 | 65
Number analyzed (Eyes) | 110 | 110
logMAR | 0.143 (0.1084) | 0.143 (0.1117)
Statistical Analysis 1: Comparison: Delefilcon A; Test type: Superiority — Statistical superiority was concluded if the upper limit of the confidence intervals of the Test lens was below +0.17 logMAR for near; Linear mixed model analysis; Linear mixed model using the Kenward and Roger method for the denominator degrees of freedom; LS Mean Estimate = 0.141, 95% CI 2-sided [0.112 to 0.170], Standard Error of Mean 0.0147
Statistical Analysis 2: Comparison: Nesofilcon A; Test type: Superiority — [test comment as in outcome 2, analysis 1]; Linear mixed model analysis; Linear mixed model using the Kenward and Roger method for the denominator degrees of freedom; LS Mean Estimate = 0.141, 95% CI 2-sided [0.112 to 0.170], Standard Error of Mean 0.0147

3. Secondary Outcome: Overall Quality of Vision
Description: Overall quality of vision was assessed using the Contact Lens User Experience™ (CLUE) questionnaire. CLUE is a validated patient-reported outcomes (PRO) questionnaire to assess patient experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120.
Time Frame: 1-Week Follow-up
Population: Subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Delefilcon A | Nesofilcon A
Number analyzed (Participants) | 65 | 65
Units on a scale | 47.4 (17.81) | 49.3 (19.43)
Statistical Analysis 1: Comparison: Delefilcon A; Test type: Superiority — Statistical superiority was concluded if the lower limit of the confidence intervals of the Test lens was above 32 CLUE points; Linear Mixed Model Analysis; Linear mixed model using the Kenward and Roger method for the denominator degrees of freedom; LS Mean Estimate = 45.5, 95% CI 2-sided [41.2 to 49.9], Standard Error of Mean 2.19
Statistical Analysis 2: Comparison: Nesofilcon A; Test type: Superiority — [test comment as in outcome 3, analysis 1]; Linear Mixed Model Analysis; Linear mixed model using the Kenward and Roger method for the denominator degrees of freedom; LS Mean Estimate = 46.4, 95% CI 2-sided [42.1 to 50.8], Standard Error of Mean 2.21

ADVERSE EVENTS:
Time Frame: Throughout the entire duration of the study. Approximately 1 month per subject.
Arm/Group | Delefilcon A | Nesofilcon A
All-Cause Mortality (participants affected / at risk) | 0/78 | 0/78
Serious Adverse Events (participants affected / at risk) | 0/78 | 0/78
Other Adverse Events (participants affected / at risk) | 0/78 | 0/78

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-01): https://cdn.clinicaltrials.gov/large-docs/23/NCT03322423/Prot_SAP_000.pdf